CLINICAL TRIAL: NCT01784016
Title: Concurrent PET D2/D3 Receptor Imaging and fMRI Smoking Cue Reactivity in Smokers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Technical complications.
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Marc J. Kaufman, Director, Translational Imaging Laboratory, McLean Hospital, Mclean Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SmokingPETD2-3fMRI; R21DA031925-01A1 (NIH)
Record Dates: First submitted 2013-01-30; First posted 2013-02-05 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Nicotine Dependence; Smoking Cue Reactivity; Relapse to Smoking
MeSH Terms: conditions — Tobacco Use Disorder | interventions — naxagolide

ARMS (2):
- Healthy Smokers (Experimental): Healthy smokers aged 18-50 years reporting average cigarette consumption of 15 or more cigarettes/day for the past year, providing an expired breath carbon monoxide reading exceeding 10 ppm at screening.
  Interventions: Radiation: [11C]-PHNO
- Healthy Nonsmokers (Experimental): Healthy nonsmoking controls aged 18-50 reporting consumption of <100 cigarettes in their lifetime, none in the last 6 months, providing an exhaled breath carbon monoxide reading of < 9 ppm at screening.
  Interventions: Radiation: [11C]-PHNO

INTERVENTIONS:
Radiation: [11C]-PHNO — [11C]-PHNO will be administered once intravenously to conduct Positron Emission Tomography (PET) measurements of dopamine D2/D3 binding potential.
  Other Names: 11C-(+)-4-propyl-3,4,4a,5,6,10b-hexahydro-2H-naphtho[1,2-b][1,4]oxazin-9-ol

SUMMARY:
This trial aims to determine whether dopamine D3 receptors are elevated in smokers versus nonsmokers and whether correlations exist between D3 receptor binding potential (BP) and functional MRI (fMRI) reactivity to smoking cues, which has been associated with smoking relapse vulnerability.

Neuroimaging measures of D3 BP and smoking cue fMRI reactivity will be collected concurrently in otherwise healthy nicotine-dependent smokers and age-matched nonsmokers using a 3 Tesla MRI scanner configured to conduct fMRI and Positron Emission Tomography (PET).

We will measure D3 receptor BP using radiolabeled [11C]-(+)-PHNO, which has a relatively higher affinity for D3 versus D2 receptors.

We hypothesize that D3 BP will be elevated in smokers versus nonsmokers and that in smokers, there will be a positive correlation between smoking cue fMRI reactivity and D3 BP.

ELIGIBILITY:
Inclusion Criteria:

* competent to provide written informed consent
* Smokers: self-report of smoking 15 or more cigarettes/day for the past year, self-report of smoking first cigarette of the day within 30 minutes of awakening, meets DSM-IV criteria for Nicotine Dependence, provides expired breath carbon monoxide reading of > 10 ppm at enrollment
* Nonsmokers: self-report of consuming <100 cigarettes in their lifetime, none in the last 6 months, provides expired breath carbon monoxide reading of < 9 ppm at enrollment
* Women of childbearing potential: negative STAT serum beta-human chorionic gonadotrophin pregnancy test before scanning

Exclusion Criteria:

* pregnant or able to become pregnant and not willing to undergo blood pregnancy test
* unstable medical illness with likely hospitalization for treatment within 6 months
* life-threatening arrhythmia, cerebro-vascular or cardiovascular event within 6 months of enrollment; liver function tests elevated over 2.5x normal; CNS tumor or seizure disorder
* users of other tobacco- or nicotine-containing products (gum, patches, e-cigarettes)
* lifetime history of DSM-IV bulimia, organic mental disorder, brain injury or psychotic disorder
* 6 month history of non-nicotine substance use disorder or major depression
* history of multiple adverse drug reactions
* current use of excluded concomitant medications (smoking cessation medications)
* known history of allergic reaction to the PET ligand [11C]-PHNO, its components, or any medication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Dopamine D3 Receptor Binding Potential Difference Between Smokers and Nonsmokers | March 2014
  We will determine whether dopamine D3 receptor binding potential, a dimensionless number which represents the relative concentration of dopamine D3 receptors available for binding, is elevated in smokers versus nonsmoking controls.

SECONDARY OUTCOMES:
Smoking Cue fMRI Reactivity Association with Dopamine D3 Receptor Binding Potential | March 2014
  In smokers, we will determine whether an association exists between smoking cue fMRI reactivity intensity (beta weight) and dopamine D3 receptor binding potential, a relationship between receptor (D3) density and dopamine occupancy.

CONTACTS AND LOCATIONS:
Overall Officials: Marc J. Kaufman, Ph.D., Principal Investigator — Mclean Hospital
Locations (3):
- United States (3):
  - McLean Hospital, Belmont, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Athinoula A. Martinos Center for Biomedical Imaging, Charlestown, Massachusetts

REFERENCES:
- [Background] Janes AC, Pizzagalli DA, Richardt S, deB Frederick B, Chuzi S, Pachas G, Culhane MA, Holmes AJ, Fava M, Evins AE, Kaufman MJ. Brain reactivity to smoking cues prior to smoking cessation predicts ability to maintain tobacco abstinence. Biol Psychiatry. 2010 Apr 15;67(8):722-9. doi: 10.1016/j.biopsych.2009.12.034. Epub 2010 Feb 20. PMID 20172508
- [Background] Le Foll B, Diaz J, Sokoloff P. Increased dopamine D3 receptor expression accompanying behavioral sensitization to nicotine in rats. Synapse. 2003 Mar;47(3):176-83. doi: 10.1002/syn.10170. PMID 12494400
- [Background] Searle G, Beaver JD, Comley RA, Bani M, Tziortzi A, Slifstein M, Mugnaini M, Griffante C, Wilson AA, Merlo-Pich E, Houle S, Gunn R, Rabiner EA, Laruelle M. Imaging dopamine D3 receptors in the human brain with positron emission tomography, [11C]PHNO, and a selective D3 receptor antagonist. Biol Psychiatry. 2010 Aug 15;68(4):392-9. doi: 10.1016/j.biopsych.2010.04.038. PMID 20599188
- [Background] Tziortzi AC, Searle GE, Tzimopoulou S, Salinas C, Beaver JD, Jenkinson M, Laruelle M, Rabiner EA, Gunn RN. Imaging dopamine receptors in humans with [11C]-(+)-PHNO: dissection of D3 signal and anatomy. Neuroimage. 2011 Jan 1;54(1):264-77. doi: 10.1016/j.neuroimage.2010.06.044. Epub 2010 Jun 30. PMID 20600980
- [Background] Wilson AA, McCormick P, Kapur S, Willeit M, Garcia A, Hussey D, Houle S, Seeman P, Ginovart N. Radiosynthesis and evaluation of [11C]-(+)-4-propyl-3,4,4a,5,6,10b-hexahydro-2H-naphtho[1,2-b][1,4]oxazin-9-ol as a potential radiotracer for in vivo imaging of the dopamine D2 high-affinity state with positron emission tomography. J Med Chem. 2005 Jun 16;48(12):4153-60. doi: 10.1021/jm050155n. PMID 15943487
- [Background] Pak AC, Ashby CR Jr, Heidbreder CA, Pilla M, Gilbert J, Xi ZX, Gardner EL. The selective dopamine D3 receptor antagonist SB-277011A reduces nicotine-enhanced brain reward and nicotine-paired environmental cue functions. Int J Neuropsychopharmacol. 2006 Oct;9(5):585-602. doi: 10.1017/S1461145706006560. Epub 2006 Aug 31. PMID 16942635